CLINICAL TRIAL: NCT07372352
Title: Clinical Study on the Efficacy and Safety of Zeprumetostat, Azacitidine Combined With Mitoxantrone Hydrochloride Liposome in Relapsed/Refractory Peripheral T-Cell Lymphoma.
Brief Title: Zeprumetostat, Azacitidine Combined With Lipo-MIT in R/R PTCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20251196
Record Dates: First submitted 2026-01-03; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Peripheral T Cells Lymphoma (PTCL)
MeSH Terms: interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zeprumetostat + Azacitidine + Lipo-MIT. (Experimental): This single-arm, Phase II study evaluates a combination regimen followed by monotherapy maintenance. All participants receive up to six 21-day cycles of induction therapy: Zeprumetostat (350 mg orally twice daily continuously), Azacitidine (100 mg subcutaneous injection on days 1-5), and Mitoxantrone Hydrochloride Liposome(Lipo-MIT) (16 mg/m² IV on day 1). Response is formally assessed after Cycle 3. Only patients achieving a Complete Response (CR) or Partial Response (PR) proceed to complete Cycles 4-6. Patients with CR or PR after induction then enter a maintenance phase of up to 2 years with Zeprumetostat monotherapy (350 mg orally twice daily). Treatment continues until disease progression, unacceptable toxicity, withdrawal of consent, or completion of the maintenance period. Protocol-defined dose modifications are permitted for adverse events.
  Interventions: Drug: Zeprumetostat; Drug: Azacitidine (AZA); Drug: Mitoxantrone Hydrochloride Liposome

INTERVENTIONS:
Drug: Zeprumetostat — Zeprumetostat is an oral, selective Enhancer of Zeste Homolog 2 (EZH2) inhibitor. EZH2 is a histone methyltransferase often dysregulated in lymphomas. By inhibiting EZH2, zeprumetostat modulates epigenetic programming to reverse aberrant gene silencing, induce cell cycle arrest and apoptosis. In this study, it is administered at 350 mg orally twice daily continuously. It is used both in the 6-cycle induction combination phase and as monotherapy in the up to 2-year maintenance phase for responding patients.
Drug: Azacitidine (AZA) — Azacitidine is a DNA methyltransferase inhibitor (hypomethylating agent). As a cytidine analog, it incorporates into DNA and RNA, leading to DNA hypomethylation, reactivation of silenced tumor suppressor genes, and direct cytotoxicity. In this study, azacitidine is administered at 100 mg via subcutaneous injection once daily on Days 1-5 of each 21-day induction cycle. It is part of the initial triple-drug induction regimen and is not used during the subsequent maintenance phase.
Drug: Mitoxantrone Hydrochloride Liposome — Mitoxantrone Hydrochloride Liposome is a liposomal formulation of the anthracenedione chemotherapy agent mitoxantrone. The liposomal encapsulation aims to improve pharmacokinetics and tissue distribution. Its mechanism involves intercalating into DNA and inhibiting topoisomerase II, causing DNA strand breaks and cell death. In this study, it is administered intravenously at 16 mg/m² on Day 1 of each 21-day induction cycle. It is used only in the initial 6-cycle combination induction phase.

SUMMARY:
This clinical trial is a Phase II study investigating the effectiveness and safety of a three-drug combination-Zeprumetostat, Azacitidine, and Mitoxantrone Hydrochloride Liposome-in adults with relapsed or refractory peripheral T-cell lymphoma (PTCL). PTCL is an aggressive type of non-Hodgkin lymphoma that has limited treatment options after the first line of therapy.

The study aims to enroll approximately 26 patients at a single center in China. Eligible participants will receive up to 6 cycles of induction therapy with all three drugs, followed by up to 2 years of maintenance therapy with Zeprumetostat alone if they respond to treatment.

The main goal is to evaluate the overall response rate (how many patients experience tumor shrinkage). Secondary goals include assessing how long patients live without their disease getting worse, how long they survive overall, and the safety profile of this treatment combination. The study will also explore whether specific genetic markers or viral infections are linked to how well patients respond.

This study is important because it tests a novel, potentially less toxic, and more effective combination for a patient population with high unmet medical need. All participants will be closely monitored for treatment response and side effects throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory peripheral T-cell lymphoma after first-line or higher treatment.
2. Age ≥ 18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 2.
4. Presence of measurable target lesions [Note: Target lesions are defined as lesions with at least one longest diameter (LD) measurement > 1.5 cm and longest perpendicular diameter (LPD) measurement ≥ 1.0 cm, as assessed by computed tomography (CT) or magnetic resonance imaging (MRI). A maximum of six target lesions can be selected].
5. Adequate function of major organs must meet the following criteria:

   * Hematological parameters: HB ≥ 70 g/L, PLT ≥ 50 × 10^9/L, NE ≥ 1.0 × 10^9/L (Note: Patients who have not received transfusions or drugs to support NE, PLT, or HB increase within 1 week before screening are eligible. Patients with bone marrow involvement by lymphoma resulting in cytopenia are not restricted by this criterion).
   * Echocardiographic left ventricular ejection fraction ≥ 50%.
   * Creatinine ≤ 132 umol/L or creatinine clearance ≥ 60 ml/min.
   * ALT and AST ≤ 3 times the upper limit of normal.
6. Women of childbearing potential must have a negative pregnancy test. Both male and female patients must agree to use effective contraception during treatment and for 1 year thereafter.
7. Life expectancy of more than 3 months.
8. Voluntary signed informed consent form.

Exclusion Criteria:

1. Underwent major surgery or severe trauma within 2 weeks before enrollment, or significant adverse effects have not yet recovered.
2. Currently suffering from or having had other malignancies within 3 years before enrollment, except for cured basal or squamous cell carcinoma of the skin, superficial bladder cancer, prostatic intraepithelial neoplasia, and cervical carcinoma in situ.
3. History of stroke or intracranial hemorrhage within the past 3 months.
4. Presence of complications or medical conditions that may interfere with the conduct of the study or pose a significant risk to the patient, including but not limited to severe cardiovascular diseases (e.g., cardiac disease classified as New York Heart Association class III or IV, myocardial infarction within the past 6 months, unstable arrhythmias, or unstable angina) and/or severe pulmonary diseases (e.g., severe obstructive pulmonary disease and history of symptomatic bronchospasm).
5. Human immunodeficiency virus infection, or presence of uncontrollable active hepatitis C virus or hepatitis B virus infection.
6. Uncontrollable active infection.
7. Pregnant or breastfeeding women.
8. Any life-threatening disease, medical condition, or organ system dysfunction that may endanger the safety of the patient, as determined by the investigator.
9. Any condition that may interfere with the absorption or metabolism of zemtovistat, azacitidine, or doneda, or place the study results at unnecessary risk.
10. Lymphoma involvement of the central nervous system.
11. Presence of conditions judged by the investigator to interfere with full participation in the study; conditions posing significant risk to the subject; or conditions that may interfere with the interpretation of study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-01-15 (Estimated); Study Completion 2029-07-15 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) after 6 treatment cycles | Efficacy will be assessed at the end of the induction therapy (6 cycles in total). Each treatment cycle is 21 days.
  The proportion of participants who achieve a Complete Response (CR) or Partial Response (PR) per the Lugano 2014 classification.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From the first dose of study treatment until the date of first documented disease progression or death from any cause, whichever occurs first, assessed up to 60 months.
Complete Response (CR) Rate after 6 treatment cycles | Efficacy will be assessed at the end of induction therapy (6 cycles in total). Each treatment cycle is 21 days.
Duration of Response (DOR) | From the date of first documented response (partial or complete) until the date of first documented disease progression or death from any cause, whichever occurs first, assessed up to 60 months.
Overall Survival (OS) | From the first dose of study treatment until the date of first documented disease progression or death from any cause, whichever occurs first, assessed up to 60 months.
Incidence of Treatment-Emergent Adverse Events (Safety) | From the first dose of study treatment until 30 days after the last dose, or until the start of new anti-cancer therapy, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No